CLINICAL TRIAL: NCT01998061
Title: Phase II Study of Continuation of Tyrosine Kinase Inhibitor (TKI) With or Without Chemotherapy Beyond Gradual Progression in Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Continuation of TKI With or Without Chemotherapy Beyond Gradual Progression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangU
Record Dates: First submitted 2013-11-24; First posted 2013-11-28 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — EGFR tyrosine kinase inhibitor 324674; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): TKI alone until rapid progression
  Interventions: Drug: EGFR tyrosine kinase inhibitor
- Arm B (Experimental): TKI combined with investigator's choice of chemotherapy regimen and subsequent line of treatment until rapid progression.
  Interventions: Drug: EGFR tyrosine kinase inhibitor with chemotherapy

INTERVENTIONS:
Drug: EGFR tyrosine kinase inhibitor — Arm A
  Other Names: EGFR TKI
  Arms: Arm A
Drug: EGFR tyrosine kinase inhibitor with chemotherapy — Arm B
  Other Names: EGFR TKI with chemotherapy
  Arms: Arm B

SUMMARY:
There have been reports suggesting that continuous administration of epidermal growth factor receptor-tyrosine kinase inhibitors (EGFR-TKIs) is advantageous for patients in which gradual disease progression was observed after the establishment of clinical benefit from EGFR-TKIs. However, whether EGFR TKI with or without chemotherapy provides more survival benefit has not been formally evaluated.

DETAILED DESCRIPTION:
We design this clinical trial to compare the efficacy of continuation of EGFR TKI with or without chemotherapy in patients beyond gradual progression.

ELIGIBILITY:
Inclusion criteria:

Patient who was confirmed stage IV NSCLC by pathologic histology or cytology. Males or females aged ≥18 years, < 75 years. Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Life expectancy ≥12 weeks.

Males and females should be contraceptive during the period of the trial until 8 weeks after the last administration of the drug.

Definition of gradual progression:

1. Slow PD (6 months of partial response/stable disease),
2. Asymptomatic minimal PD,
3. New brain metastasis controlled locally. Patients with asymptomatic, treated brain metastases are eligible for trial participation.

Adequate bone marrow, renal, and liver function are required. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Institutional review board-approved informed consent will be obtained for every patient before initiation of any trial-specific procedure or treatment.

Exclusion criteria： Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).

Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.

Female subjects should not be pregnant or breast-feeding. Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.

Adequate renal function: Serum creatinine ≤ 1.5 x ULN, or ≥ 50 ml/min. Adequate liver function :Total bilirubin £ 1.5 x upper limit of normal (ULN) and Alanine Aminotransferase (ALT )and Aspartate Aminotransferase (AST )< 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.

Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 18 months

SECONDARY OUTCOMES:
Objective response rate cacy | up to 18 months

OTHER OUTCOMES:
Quality of life | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qiong Zhao, Hangzhou, Zhejiang, China